CLINICAL TRIAL: NCT04584827
Title: Evaluation of Lactate in Patients Undergoing Glial and Non Glial Mass Surgery With Craniotomy
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Onur Kucuk, Department of anesthesiology and reanimation, Research Assistant, Trakya University
Other Study IDs: TÜTF-BAEK 2019/450
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Lactate; Brain Tumor; Post-Op Complication
Keywords: lactate; glial and non glial tumor; intracranial; craniotomy
MeSH Terms: conditions — Brain Neoplasms; Postoperative Complications | interventions — Lactase; Glasgow Outcome Scale

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- complication positive (up to 30 days after surgery): Complications:
  * Moderate to severe intracerebral hemorrhage confirmed in a brain CT scan (Midline shift in brain imaging ≥ 3 mm),
  * İntracranial hypertension requiring post op surgical drainage,
  * Status epilepticus or seizures,
  * The need for tracheal intubation or use of mechanical ventilation after surgery,
  * Decrease in GKS,
  * Unmanageable agitation that requires restriction or sedation,
  * Need for respiratory failure and oxygen therapy,
  * Unexpected serious motor deficit
  * Died
  Interventions: Other: lactate level; Other: Glasgow Outcome Scale
- complication negative (up to 30 days after surgery): No complications are seen within 30 days and the patient is healthy
  Interventions: Other: lactate level; Other: Glasgow Outcome Scale

INTERVENTIONS:
Other: lactate level — Lactate, a byproduct of glycolysis, is an indicator of weak tissue perfusion and a useful biomarker with prognostic value in various diseases. Lactate value is calculated by blood gas.
  Other Names: lac
Other: Glasgow Outcome Scale — Glasgow Outcome Scale; It is a scale developed to categorize people suffering from head trauma or non-traumatic acute brain injury into broad outcome categories. It shows postoperative mortality and morbidity of patients who underwent intracranial surgery.
  Other Names: GOS

SUMMARY:
The aim of this study is to determine the effects of the level of metabolites used in routine on mortality and morbidity in patients who will undergo intracranial surgery with craniotomy.

DETAILED DESCRIPTION:
In this study, in patients who are planned to have an intracranial mass operation with craniotomy, their medical histories, demographic features, comorbidities, preoperative radiotherapy treatment, the parameters examined in the preoperative routine will be collected as a file scan (previous operations, GKS, laboratory values). The classification of patients according to the 2016 World Health Organization Central Classification of Nervous System Tumors (WHO-CNS classification) and whether it is glial or non glial will be recorded from the clinical file. Intraoperative; hemodynamic data of patients; heart rate, diastolic, systolic and mean arterial pressures, fluid and blood products delivered, anesthetic and other medications, and blood gas samples will be written from the anesthesia document after the operation is finished. For the study, the application of the anesthesiologist for the patient will not be interfered. If postoperative patients are sent to the intensive care unit, their laboratory values and clinical observations (mortality, morbidity, neurological sequelae, imaging techniques, GOSE (Glasgow outcome skale)) will be recorded. In our study, mortality and morbidity will be evaluated 30 days postoperatively, and if the patient was sent to the service from the intensive care unit in this process, the values in the postoperative clinic (mortality, morbidity, neurological evaluation, imaging techniques, pathology results) will be recorded from the patient document. If the patient was discharged 30 days before, outpatient data will be recorded. The patients will be classified by evaluating the collected data (intraoperative hemodynamic data, blood transfusions, postoperative neurological sequel, postoperative complications and mortality).

In our study; the effects of lactate level on mortality and morbidity will be investigated in patients undergoing an intracranial mass operation with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Having an intracranial mass operation with craniotomy
2. No history of congestive heart failure
3. No kidney and liver dysfunction
4. Not pregnant
5. Not taking inotropic drugs during the operation
6. Receiving less than four red blood product replacements during the operation

Exclusion Criteria:

1. Patients with a history of congestive heart failure
2. Patients with kidney and liver dysfunction
3. Patients who need an inotropic agent to adjust blood pressure during the operation
4. Patients who have undergone four or more red blood product transfusions during the operation
5. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to include intracranial mass operations performed by craniotomy between 10 December 2019 - 10 December 2020 in Trakya University Faculty of Medicine, Department of Neurosurgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
lactate level | change from operation to post-op second day (4 time)
  Lactate, a byproduct of glycolysis, is an indicator of weak tissue perfusion and a useful biomarker with prognostic value in various diseases. Lactate value is calculated by blood gas.

SECONDARY OUTCOMES:
Glasgow Outcome Scale | 30 days after the operation (1 time)
  Glasgow Outcome Scale; It is a scale developed to categorize people suffering from head trauma or non-traumatic acute brain injury into broad outcome categories. It shows postoperative mortality and morbidity of patients who underwent intracranial surgery. Glasgow Outcome Scale is a five-point scale. 1 point is considered death and five points as good recovery. As the score increases, morbidity and mortality decrease.

CONTACTS AND LOCATIONS:
Overall Officials: SEVTAP HEKİMOĞLU ŞAHİN, Professor, Principal Investigator — Trakya University; ONUR KÜÇÜK, Resident, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Centrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No